CLINICAL TRIAL: NCT02812394
Title: A Phase 1 Single Dose Pharmacokinetic Bridging Study to Compare Two Dose Strengths of CVT-301 (Levodopa Inhalation Powder) With an Oral Dose of Sinemet® (Carbidopa-levodopa) Tablets
Brief Title: A Study to Compare Two Dose Strengths of CVT-301 (Levodopa Inhalation Powder) With an Oral Dose of Sinemet® (Carbidopa-levodopa) Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Acorda Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVT-301-010
Record Dates: First submitted 2016-06-22; First posted 2016-06-24 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; Episodic motor fluctuations (OFF periods)
MeSH Terms: conditions — Parkinson Disease | interventions — carbidopa, levodopa drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CVT-301 (Experimental): CVT-301 (Dose Level 1): two (low dose) levodopa fine particle dose (FPD) capsules administered to the lung via oral inhalation using the CVT 301 inhaler.
  CVT-301 (Dose Level 2): two (high dose) levodopa FPD capsules administered to the lung via oral inhalation using the CVT 301 inhaler.
  Sinemet® (carbidopa/levodopa)
  Interventions: Drug: CVT-301 (Dose Level 1); Drug: CVT-301 (Dose Level 2); Drug: Sinemet®

INTERVENTIONS:
Drug: CVT-301 (Dose Level 1) — All subjects will receive a single dose of low-dose CVT-301 with a 1-day washout between the doses.
Drug: CVT-301 (Dose Level 2) — All subjects will receive a single dose of high-dose CVT-301 with a 1-day washout between the doses.
Drug: Sinemet® — All subjects will receive carbidopa/levodopa tablets administered every 8 hours.
  Other Names: carbidopa/levodopa

SUMMARY:
This study will be an open-label, randomized, three-period cross-over pharmacokinetic evaluation of CVT-301 compared with the Reference Listed Drug (RLD), orally administered carbidopa/levodopa, in healthy volunteers.

DETAILED DESCRIPTION:
The primary objective is to determine the relative bioavailability of two CVT-301 (dose levels 1 and 2) capsules compared with the Reference Listed Drug (RLD) on a per milligram basis.

ELIGIBILITY:
Inclusion Criteria:

* In good general health as determined by medical history, physical examination, electrocardiogram (ECG), vital signs, and clinical laboratory evaluation;
* FEV1/FVC above the 5th percentile of the predicted normal distribution for age and gender;
* Body Mass Index (BMI) between 18 - 30 kg/m2

Exclusion Criteria:

* No flu-like syndrome or other respiratory infections within 2 weeks prior to the Screening Visit;
* Negative drug and alcohol testing;
* Negative pregnancy test for female subjects

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-06; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma drug concentration (Cmax) | within 15min pre-dose (baseline) and specified time points up to and @ 24h post-dose.
Area under the plasma concentration curve from time 0 to the concentration at 24 hours (AUC0-24h) | within 15min pre-dose (baseline) and specified time points up to and @ 24h post-dose.

SECONDARY OUTCOMES:
Number of subjects with Adverse Events (AEs) including Serious AEs | up to 9 days

CONTACTS AND LOCATIONS:
Overall Officials: Charles Oh, MD, Study Director — Acorda Therapeutics
Locations (1):
- Site #001, Dallas, Texas, United States